CLINICAL TRIAL: NCT00948662
Title: Ascending Single Dose Study Of The Safety, Tolerability And Pharmacokinetics Of SAM-760 Administered Orally To Healthy Young And Healthy Elderly Subjects
Brief Title: Study Evaluating The Safety And Tolerability Of Administration Of Single Oral Doses Of SAM-760 To Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3276A1-1000; B2081001; NCT01298453 (obsolete NCT alias)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Safety; tolerability; ascending single doses; healthy subjects
MeSH Terms: interventions — SAM-760; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): active arm/healthy young
  Interventions: Drug: SAM-760
- 2 (Placebo Comparator): placebo arm
  Interventions: Drug: Placebo of SAM-760
- 3 (Other): ketoconazole interaction evaluation
  Interventions: Drug: ketoconazole

INTERVENTIONS:
Drug: SAM-760 — SAM-760 capsule, 0.25, 0.75, 2.25, 5, 10, 15, 20, 25, 35 and 45mg, single dose, 1 day
  Arms: 1
Drug: Placebo of SAM-760 — SAM-760 matching placebo capsule, single dose, 1 day,
  Other Names: Placebo
  Arms: 2
Drug: ketoconazole — Ketoconazole oral tablets, 200 mg bid, 14 days
  Other Names: ketoconazole interaction arm
  Arms: 3

SUMMARY:
This study will assess the safety and tolerability of ascending single oral doses of SAM-760 in healthy young adult and healthy elderly subjects. The secondary objectives are to provide the concentrations of SAM-760 in the blood and to evaluate the effect of a high-fat meal on the concentrations in the blood of SAM-760 administered to healthy young adult subjects, and to evaluate the effects of concomitant administration of ketoconazole on the safety and the concentrations of SAM-760 in the blood of a single dose of SAM-760 in healthy young adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential aged 18 to 50 years inclusive (healthy young subjects) and > 65 years (healthy elderly subjects) at screening.
* Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight >= 50 kg.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the investigational drug or placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 5 days

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for PF-05212377 over time. | 5 days
Measurement of Area Under the curve (AUC) for PF-05212377. | 5 days
Time of maximum (Tmax) concentration of PF-05212377 in plasma. | 5 days
Elimination half life (t1/2) of PF-05212377. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Rueil-Malmaison, France, France

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3276A1-1000&StudyName=Study%20Evaluating%20The%20Safety%20And%20Tolerability%20Of%20Administration%20Of%20Single%20Oral%20Doses%20Of%20SAM-760%20%20To%20Healthy%20Subjects